CLINICAL TRIAL: NCT07098845
Title: Testing a Mindfulness-Based Intervention With a Multi-Modal Adaptive Supplement for Stress-Related Problems in College Students
Brief Title: Mindfulness-Based Intervention With a Supplement for Stress-Related Problems in College Students Across Multiple Sites (4SITE)
Acronym: 4SITE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: University of Minnesota (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH); University of Colorado, Denver (Other); Macalester College (Unknown)
Responsible Party: Principal Investigator, Rachel Graham, Professor of Human Development & Family Studies and Colorado School of Public Health, Colorado State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 5036; 1R01AT012652 (NIH)
Record Dates: First submitted 2025-06-10; First posted 2025-08-01 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Stress; Mental Health; Mindfulness Based Stress Reduction
Keywords: Mindfulness; Stress; College Students; Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Learning to BREATHE (L2B) (Active Comparator)
  Interventions: Behavioral: Learning to BREATHE
- Learning to BREATHE Plus (L2B PLUS) (Experimental)
  Interventions: Behavioral: Learning to BREATHE Plus
- HealthEd (Active Comparator)
  Interventions: Behavioral: HealthEd

INTERVENTIONS:
Behavioral: Learning to BREATHE — L2B is a group MBI designed for adolescents (Broderick & Metz, 2009) and teaches three families of practices: focused attention (e.g., breath awareness), open awareness (i.e., awareness of sensations, thoughts, and feelings as they occur), and compassion. Each letter in BREATHE corresponds to a theme: Body, Reflections, Emotions, Attention, Tenderness, and Habits, building to the overall goal of Empowerment. Each session involves guided discussions, activities, and mindfulness practices.
  Other Names: L2B
  Arms: Learning to BREATHE (L2B)
Behavioral: Learning to BREATHE Plus — The in-person, group program portion of L2B PLUS and L2B are identical. But, L2B PLUS (Lucas-Thompson et al., 2020) builds on the standard L2B program with 3 additional supplements: 1) Extensive on-demand library designed by the team to be integrated with the group program and specifically to allow participants to independently practice skills that have already been introduced in the group program. 2) Intervention messages sent across the day. The team developed intervention messages to be sent 5 times a day to participants (Lucas-Thompson et al., 2020). Each week, participants receive intervention content tailored to what they have just learned in the group program. 3) JIT support. When participants indicate high stress via EMAs completed during the intervention period, tailored intervention content is delivered "just-in-time" during a moment of high need. These JIT messages were developed specifically to support applying or using mindfulness during periods of high stress.
  Other Names: L2B PLUS
  Arms: Learning to BREATHE Plus (L2B PLUS)
Behavioral: HealthEd — Hey-Durham is a health education program that the team has extensive experience implementing (Lucas-Thompson et al., 2019; Shomaker, Berman, et al., 2019; Shomaker et al., 2016; Tanofsky-Kraff et al., 2014) and covers topics such as domestic violence, substance use, depression/signs of suicide, and conflict resolution. Mental health components focus only on prevalence and identification. There is no content overlap with L2B, but it is matched to L2B in format, time, frequency, in-person contact, and facilitator expertise. Inclusion of HealthEd in a future efficacy trial will allow us to test the extent to which the active ingredients of MBI (i.e,. a top-down and bottom-up focus on emotion and stress regulation(Zelazo & Carlson, 2012)), with and without the between-session support L2B, improve mental health and stress responding, relative to an active control matched for critical characteristics but that does not include these active ingredients.
  Other Names: Hey-Durham
  Arms: HealthEd

SUMMARY:
The investigators hope to add to the feasible, acceptable, and effective interventions that offer reductions in depression, anxiety, and stress for students at U.S. colleges and universities, the majority of whom experience mental health problems but the minority of whom who receive adequate mental health support. By studying the extent to which a multi-modal supplement boosts effects for a mindfulness-based intervention (and comparing both to an active health education control program) to reduce depression, anxiety, and stress, the proposed research seeks to rigorously investigate complementary and integrative health interventions and their roles in improving health.

DETAILED DESCRIPTION:
There have been dramatic and concerning increases in rates of psychological distress in students enrolled in US colleges and universities over the last decade. The majority of college students in the last year experienced mental health problems, and if left untreated, symptoms of these problems have serious individual and public health consequences, both in the short- and long-term. However the vast majority of students do not receive professional mental health support because traditional treatments are perceived as ineffective and inconvenient. Additionally, many on campus resources cannot meet the demand of students needing support. As a result, it is critical to identify acceptable and effective interventions to address what is being called a "campus mental health crisis." Mindfulness-based interventions (MBIs) are very well-liked by college students, most of whom are late adolescents; in addition they are effective at increasing mindfulness and emotion regulation as well as reducing stress and depression. However, MBI effects have typically been small-to-moderate. Outside of the mindfulness literature, technological supplements to group-based programs like MBIs have been found to be effective at increasing intervention efficacy. The investigative team developed the first multi-modal adaptive supplement to an MBI (5K01AT009592), Learning To BREATHE PLUS ( L2B PLUS), which supplements an evidence-based group MBI with multiple methods of support for practicing mindfulness in daily life. The investigators program of research provides evidence at a single site that L2P PLUS is feasible and highly acceptable to adolescents, results in sustained levels of engagement across the group program period, and appears to be more effective than the standard Learning To BREATHE group program (L2B) at increasing daily mindfulness practice and consistency of mindfulness during stress as well as reducing psychological distress. In turn, L2B appears more effective in reducing stress-related behavior compared to an active, didactic health education control (HealthEd). Building directly on the investigators' prior work the proposed R01 study is a multisite, pilot randomized controlled trial implemented at four sites in order to prepare for a future multi-site efficacy trial testing the effects of L2B PLUS relative to the standard L2B program and HealthEd on depression, anxiety, and stress. Specific aims of the current proposal are to: 1) evaluate multi-site fidelity of training and implementation of 6-week L2B PLUS, 6 week L2B and 6-week HealthEd to college students experiencing stress, 2) test multi-site feasibility and acceptability of recruitment, retention, and protocol adherence for randomized control trial (RCT) involving L2B PLUS, L2B, and HealthEd, and 3) modify training/implementation and protocol for a future, fully powered multi-site efficacy trial. Completion of these aims will prepare us for an adequately-powered, multi-site efficacy trial, and ultimately inform a complementary and integrative approach to supporting college students experiencing problems with stress.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-25 years
* enrolled in a college or university
* experiencing elevated stress
* plan to be available in-person in the semester following the study
* own a smart phone.

Exclusion Criteria:

* have several depressive symptoms
* have suicidal ideation.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Program-specific intervention knowledge evaluations | 2 months before baseline
  Post-training L2B, L2B PLUS, and HealthEd knowledge assessments (0-25) will be completed by facilitators with higher scores indicating higher intervention knowledge
Number of eligible participants recruited with elevated stress as assessed by the Perceived Stress Scale | Within a 12-month period
  Study goal of 120 participants total across 4 sites who have elevated stress (>14) on the Perceived Stress Scale (0-40) where higher scores indicate higher stress
Program-specific facilitator adherence ratings of mock intervention group sessions | 2 months before baseline
  Facilitator adherence to each intervention manual (0-100) for L2B, L2B PLUS, and HealthEd, during mock sessions after intervention facilitation training where higher scores mean higher adherence
Program-specific facilitator competence ratings of mock intervention group sessions | 2 months before baseline
  Facilitator competence of each intervention manual (0-100) for L2B, L2B PLUS, and HealthEd, during mock sessions after intervention facilitation training where higher scores mean higher competence
Percentage of eligible students who enroll | Within a 12-month period
Percentage of enrolled participants who attend 5/6 intervention sessions | During 6-week interventions
Acceptability ratings of intervention by participants | Within one-month of intervention end
  Acceptability ratings (1-5) with higher scores meaning higher acceptability
Qualitative assessment of acceptability of interventions | Within one-month of intervention end
  Focus within group programs will qualitatively assess the acceptability of interventions
Percent of participants retained at post-test | Post intervention, 6 weeks after baseline
Percent retention at six-month follow-up | 32 weeks after baseline
Adherence to standardized data collection protocol measured via standardized checklists | At baseline, 6 weeks after, and 32 weeks after
  Percentage of data collection protocol adhered to by assessors (0-100) with higher scores indicating better adherence

SECONDARY OUTCOMES:
Depressive Symptoms | At baseline, 6 weeks after, and 32 weeks after
  Participant depressive symptoms will be assessed using the Center for Epidemiological Studies Depression Scale (Radloff, 1977). The Center for Epidemiological Studies Depression Scale has 20 questions rated on a 1-4 Likert scale where higher scores indicate higher depressive symptoms.
Clinical Depression | At baseline, 6 weeks after, and 32 weeks after
  Participant levels of clinical depression will be assessed using the Beck Depression Inventory (Beck et al., 1961). The Beck Depression Inventory has 21 questions rated on a 0-3 Likert scale where higher scores indicate higher depressive symptoms.
Anxiety | At baseline, 6 weeks after, and 32 weeks after
  Participant anxiety will be assessed using the State-Trait Anxiety Inventory (Beiling et al., 1998). It has 20 questions rated on a 1-4 Likert scale where higher scores indicate higher anxiety.
Perceived Stress | At baseline, 6 weeks after, and 32 weeks after
  Participant perceived stress will be assessed using the Perceived Stress Scale (Cohen et al., 1983). It has 14 questions rated on a 0-4 Likert scale where higher scores indicate higher perceived stress.
Social Support | At baseline, 6 weeks after, and 32 weeks after
  Participant social support will be assessed using the Multidimensional Scale of Percevied Social Support (Zimet et al., 1988). It has 12 questions rated on a 1-7 Likert scale where higher scores indicate higher social support.
Meaning in Life | At baseline, 6 weeks after, and 32 weeks after
  Participant meaning in life will be assessed using the Meaning in Life Questionaire (Steger et al., 2006). It has 10 questions rated on a 1-7 Likert scale where higher scores indicate higher meaning in life.
Mindful Attention | At baseline, 6 weeks after, and 32 weeks after
  Participant mindful attention will be assessed using the Mindful Attention and Awareness Scale (Brown et al., 2011). It has 14 questions rated on a 1-6 Likert scale where higher scores indicate higher mindful attention.
Self Compassion | At baseline, 6 weeks after, and 32 weeks after
  Participant self compassion will be assessed using the Self Compassion Scale Short Form Attention (Raes et al., 2011). It has 12 questions rated on a 1-5 Likert scale where higher scores indicate higher self compassion.
Application of Mindfulness | At baseline, 6 weeks after, and 32 weeks after
  Participant application of mindfulness will be assessed using the Applied Mindfulness Process Scale (Roemer & Medvedev, 2022). It has 15 questions rated on a 1-5 Likert scale where higher scores indicate higher mindfulness application.
Previous Experience with Mindfulness | At baseline, 6 weeks after, and 32 weeks after
  Participant previous experience with mindfulness will be assessed using the mindfulness experience and knowledge questionnaire (Qian Lau & Olivia, 2023). The mindfulness experience and knowledge questionnaire has 1 question rated on a 1-5 scale where higher scores indicate more previous mindfulness experiences.
Previous Experience with Meditation | At baseline, 6 weeks after, and 32 weeks after
  Participant previous experience with mindfulness will be assessed using a meditation questionnaire (Russell et al., 2018). The meditation questionnaire has 3 questions rated on a 1-3 Likert scale where higher scores mean more meditation knowledge.
Cortisol stress reactivity | 3 visits; baseline, after 6-week intervention, and at 6-month followup
  Cortisol reactivity to a stressor will be assessed via saliva samples collected before stressor as a test, before stressor as a baseline, immediately after stressor, and 10 minutes and 20minutes after stressor. Area under the curve will be calculated.
Blood pressure reactivity | 3 visits; baseline, after 6-week intervention, and at 6-month followup
  To assess blood pressure reactivity to a stressor, participant blood pressure will be measured at three minutes intervals across baseline and during the stressor. Change from baseline to stressor will be calculated.
Heart rate reactivity | 3 visits; baseline, after 6-week intervention, and at 6-month followup
  To assess cardiovascular reactivity to a stressor, participant heart rate will be measured at three minutes intervals across baseline and during the stressor. Change from baseline to stressor will be calculated.
Daily mindful attention | During the 6-week group program
  On a 5 question scale, with answer choices ranging from 1-6 (Brown & West, 2003), participants will report on their mindfulness each day during the group program. Higher scores indicate greater mindlessness.
Daily self-compassion | During the 6-week group program
  Participants will report their self-compassion each day during the group program using two questions (answer choices: 1 not at all to 10 extremely), with high scores indicating greater self-compassion.
Daily home practice of intervention material | During the 6-week group program
  Each day during the group program, participants will be asked to describe the extent to which the formally (1 question) and informally (1 question) engaged with what they learned in their group program (Bijkerk et al., 2023). Higher scores indicate greater engagement.
Daily negative events | During the 6-week group program
  Participants will list up to 5 negative events that occurred each day and, for each, rate their severity (from 0=not at all severe to 5=extremely severe) (Hankin et al., 2005).
Daily psychological distress | During the 6-week group program
  Each day, participants will be asked to report their psychological distress using the short-form (4 item) of the perceived stress scale (Cohen et al., 1983). Answer choices range from 1=never to 5=very often; higher scores indicate greater distress.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Lucas-Thompson, Dr., Principal Investigator — Colorado State University
Locations (4):
- United States (4):
  - University of Colorado Denver, Denver, Colorado
  - Colorado State University, Fort Collins, Colorado
  - Macalester College, Saint Paul, Minnesota
  - University of Minnesota, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No
Researchers interested in using these data to test novel hypotheses can contact the corresponding author and submit a data proposal form to be reviewed by the study team.